CLINICAL TRIAL: NCT01309360
Title: Ultrasound-guided Block of the Brachial Plexus Using Prilocaine: Effects of Local-anesthetic Dose Reduction on Parameters of Block Quality and Adverse Effects in Outpatients
Brief Title: Ultrasound-guided Axillary Plexus Block - Dose Reduction of Prilocaine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helios Research Center (Other)
Responsible Party: Dr.med. Ronald Seidel, Klinik für Anästhesiologie und Intensivtherapie, Helios Kliniken Schwerin, Wismarsche Strasse 393-7, DE-19049 Schwerin
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A 2009 24
Record Dates: First submitted 2011-03-04; First posted 2011-03-07 (Estimated); Results first posted 2011-06-27 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-06

CONDITIONS: Other Surgical Procedures
Keywords: ultrasound; methaemoglobin; prilocaine; regional anesthesia; ASA risk groups I-II; adult outpatients; surgical spectrum covered procedures; distal forearm; hand
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- group A : 40ml Prilocaine 1% (Active Comparator): 40 outpatients : 40ml Prilocaine 1% were administered for axillary plexus block
  Interventions: Drug: midazolam; Drug: prilocaine 1%
- group B : 30ml Prilocaine 1% (Active Comparator): 40 outpatients : 30ml prilocaine 1% were administered for axillary plexus block
  Interventions: Drug: midazolam; Drug: prilocaine 1%
- group C : 20ml Prilocaine 1% (Active Comparator): 40 outpatients : 20ml prilocaine 1% were administered for axillary plexus block
  Interventions: Drug: midazolam; Drug: prilocaine 1%

INTERVENTIONS:
Drug: midazolam — Prior to performing the regional anesthesia the investigators administered midazolam as a premedication by mouth (3,75-7,5mg) or intravenously (2-3mg).
  Other Names: Dormicum
Drug: prilocaine 1% — 40 outpatients : 40ml prilocaine 1% were administered for axillary plexus block
  Other Names: Xylonest 1%
  Arms: group A : 40ml Prilocaine 1%
Drug: prilocaine 1% — 40 outpatients : 30ml prilocaine 1% were administered for axillary plexus block
  Other Names: Xylonest 1%
  Arms: group B : 30ml Prilocaine 1%
Drug: prilocaine 1% — 40 outpatients : 20ml prilocaine 1% were administered for axillary plexus block
  Other Names: Xylonest 1%
  Arms: group C : 20ml Prilocaine 1%

SUMMARY:
Clinical aim: Does reducing the dose of local anesthetic in ultrasound-guided axillary plexus anesthesia have any effect on the success rate and additional parameters of block quality? Methodology: In this prospective cohort study three groups of 40 outpatients each were administered dosages of 1% prilocaine of either 40mL, 30mL or 20mL for axillary plexus anesthesia. Met-Hb was measured prior to administration of the block and then hourly until the Met-Hb concentration fell. Parameters of block quality and any adverse effects were recorded. The level of significance was defined with α ≤ 0.05.

DETAILED DESCRIPTION:
Background

With the availability of high resolution portable ultrasound equipment, the use of sonography in the field of anesthesia has become more widespread in recent years. The investigators would like to draw attention to a meta-analysis of prospective randomized studies by Abrahams et al. as being representative of the numerous publications available. Compared to nerve stimulation, ultrasound-guided nerve blocks have a higher success rate with significantly fewer vascular punctures and shorter procedure times. However, the administration of ultrasound-guided regional anesthesia necessitates considerable equipment acquisition and training expenses. Nevertheless, the suggested benefits resulting from savings in time and local anesthetic, increased patient satisfaction and avoidance of complications should be considered in addition to the results from Abrahams et al.

The aim of the present work was to investigate whether an ultrasound-guided block combined with a reduced dose of the local anesthetic prilocaine altered the success rate or other parameters of block quality. Any adverse effects and the methaemoglobin concentration were also recorded.

Methodology

After receiving ethics committee approval and after informing patients, ultrasound-guided axillary plexus anesthesia was carried out on 120 adult outpatients in ASA risk groups I-II. The surgical spectrum covered procedures on the distal forearm or the hand (carpal tunnel syndrome, ganglion extirpation, removal of material, etc.). Provision of information and inclusion in the study was done in the anesthesia outpatients' clinic as part of the standard preoperative preparation. Prior to administering the regional anesthesia the investigators administered midazolam as a premedication by mouth (3,75-7,5mg) or intravenously (2-3mg). Application of the local anesthesia was done prospectively and single blind in 3 cohorts with decreasing dosage. The patients received either 400mg (group A), 300mg (group B) or 200mg (group C) of prilocaine 1%. The block was performed under sterile conditions using a portable ultrasound device (Sonosite S-Nerve) and a 24 G short bevel cannula with flexible tubing. The block was performed using combined out-of-plane (n. musculocutaneous) and in-plane techniques (n.radialis, n.medianus, n.ulnaris), usually from a single puncture site. The outpatients were cared for in the anesthesia care unit preoperatively and postoperatively until their discharge. NIBP, pulse oxymetry and ECG were continuously monitored. The discharge criteria were widespread regression of the block with a subjective feeling of well-being including adequate analgesia and stable vital signs with methemoglobin (Met-Hb) concentrations ≤ 5%. Met-Hb levels were measured using spectrophotometry prior to the anesthesia (baseline value) and then hourly after performing the block until a clear decrease became apparent. A complete sensory block of all 4 nerves within 60 minutes of administration of the local anesthetic was rated as a successful block.

For the statistical analysis the investigators selected distribution-free, nonparametric test methods. The Mann-Whitney U test was used when comparing 2 groups and the Kruskal-Wallis test or Fisher's exact test was used when comparing more than 2 groups. The level of significance was defined with α ≤ 0.05. With multiple paired comparisons the significance level was adjusted using the Bonferroni correction. The Bravais-Pearson correlation coefficient rho describes the relationship between the maximum Met-Hb value and the weight-based prilocaine dose in mg/kg.

ELIGIBILITY:
Inclusion Criteria:

* elective surgery on the distal forearm or the hand
* adult outpatients, age 18-75 years old
* ASA-risk groups I-II (American Society of Anesthesiologists)
* Body Mass Index 17-35
* informed consent

Exclusion Criteria:

* severe coagulopathy
* local or systemic inflammatory response
* ASA-risk groups ≥ Grad III
* severe anemia
* heart failure
* manifest shock
* other drugs with influence on methaemoglobinemia (nitrates, sulfonamides etc.)
* domestic care after surgery not ensured
* drug allergy : local anesthetics
* severe polyneuropathy
* pregnancy, lactation period
* participation in other studies
* non-cooperative patients
* addiction to drugs or alcohol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Seidel, Dr. med., Principal Investigator — Klinik für Anästhesiologie und Intensivtherapie, Helios Kliniken Schwerin, Wismarsche Strasse 393-7, DE-19049 Schwerin; Georg Rehmert, Dr.med., Study Director — Klinik für Anästhesiologie und Intensivtherapie, Helios Kliniken Schwerin, Wismarsche Strasse 393-7, DE-19049 Schwerin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Provision of information and inclusion in the study was done in the anesthesia outpatients clinic as part of the standard preoperative preparation.
Pre-assignment Details: Outpatients were prematurely dropped out for medical or non-medical reasons. Non-medical reasons:1.recall of the approval by the patient, 2.unavailability of the ultrasound-machine, 3.the planned operation was not carried out. Medical reasons: severe complications like systemic toxicity of the local anesthetic (seizure, cardiac arrest).
Period: Overall Study
Arm/Group | Group A : 40ml Prilocaine 1% | Group B : 30ml Prilocaine 1% | Group C : 20ml Prilocaine 1%
Started | 40 | 40 | 40
Completed | 40 | 40 | 40
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A : 40ml Prilocaine 1% | Group B : 30ml Prilocaine 1% | Group C : 20ml Prilocaine 1% | Total
Number analyzed (Participants) | 40 | 40 | 40 | 120
Age Continuous [Mean (Standard Deviation); unit: years] | 50 (14) | 47 (16) | 45 (16) | 47 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 20 | 24 | 67
  Male | 17 | 20 | 16 | 53
percentage of methemoglobin [Mean (Standard Deviation); unit: percentage of methemoglobin] — Baseline levels of Met-Hb (percentage of methemoglobin) were measured using spectrophotometry prior to the anesthesia.
  percentage of methemoglobin | 0.84 (0.15) | 0.9 (0.16) | 0.86 (0.17) | 0.87 (0.16)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Sensory Block
Description: The number of outpatients with complete sensory block of all 4 nerves (n.musculocutaneous, n.radialis, n.ulnaris,n.medianus) was registrated in each group.
Time Frame: 60 minutes after administration of the local anesthetic
Population: The analysis was per protocol.
Measure: Number; unit: participants
Arm/Group | Group A : 40ml Prilocaine 1% | Group B : 30ml Prilocaine 1% | Group C : 20ml Prilocaine 1%
Number analyzed (Participants) | 40 | 40 | 40
participants | 38 | 39 | 39
Statistical Analysis 1: Comparison: Group A : 40ml Prilocaine 1% vs Group B : 30ml Prilocaine 1%; Test type: Superiority or Other; p = 1, Fisher Exact
Statistical Analysis 2: Comparison: Group A : 40ml Prilocaine 1% vs Group C : 20ml Prilocaine 1%; Test type: Superiority or Other; p = 1, Fisher Exact
Statistical Analysis 3: Comparison: Group B : 30ml Prilocaine 1% vs Group C : 20ml Prilocaine 1%; Test type: Superiority or Other; p = 1, Fisher Exact

2. Secondary Outcome: Maximum Concentrations of Methemoglobin
Description: Concentration of Methemoglobin (Met-Hb) was measured using spectrophotometry prior to the anesthesia (baseline value) and then hourly after performing the block until a clear decrease became apparent. The maximum amount was reached in every case two or three hours after administration of the local anesthetic.
Time Frame: 0,1,2,3,4 hours post-dose
Population: Methemoglobin (Met-Hb) levels were measured using spectrophotometry prior to the anesthesia (baseline value) and then hourly after performing the block until a clear decrease became apparent.The mean maximum Met-Hb was estimated in each group.
Measure: Mean (Standard Deviation); unit: percentage of methemoglobin
Arm/Group | Group A : 40ml Prilocaine 1% | Group B : 30ml Prilocaine 1% | Group C : 20ml Prilocaine 1%
Number analyzed (Participants) | 40 | 40 | 40
percentage of methemoglobin | 4.7 (2.1) | 3.7 (1.3) | 2.4 (0.7)
Statistical Analysis 1: Comparison: Group A : 40ml Prilocaine 1% vs Group B : 30ml Prilocaine 1% vs Group C : 20ml Prilocaine 1%; Test type: Superiority or Other; p = 0, Kruskal-Wallis

3. Secondary Outcome: Number of Participants With Objective Adverse Events as a Measure of Safety and Tolerability
Description: In groups A, B and C was determined the rate of objective clinical signs of increased Met-Hb-levels : drops in oxygen saturation <93% using pulseoximetry or lip cyanosis.
Time Frame: Outpatients were followed for the duration of hospital stay, an average of six hours.
Measure: Number; unit: participants
Arm/Group | Group A : 40ml Prilocaine 1% | Group B : 30ml Prilocaine 1% | Group C : 20ml Prilocaine 1%
Number analyzed (Participants) | 40 | 40 | 40
participants | 13 | 5 | 1
Statistical Analysis 1: Comparison: Group A : 40ml Prilocaine 1% vs Group B : 30ml Prilocaine 1%; Test type: Superiority or Other; p = 0.059, Fisher Exact
Statistical Analysis 2: Comparison: Group A : 40ml Prilocaine 1% vs Group C : 20ml Prilocaine 1%; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 3: Comparison: Group B : 30ml Prilocaine 1% vs Group C : 20ml Prilocaine 1%; Test type: Superiority or Other; p = 0.2, Fisher Exact

4. Primary Outcome: Number of Participants With Complete Motor Blocks
Description: To examine the extent of the motor block the manual muscle function test after Vladimir Janda was used. As a complete motor block was defined, when no motion (grade zero after Janda) of muscles innervated by the four blocked nerves (musculocutaneous, median, radial and ulnar nerve) was observed within 60 minutes after administration of the local anesthetic.
Time Frame: Within 60 minutes after administration of the local anesthetic
Population: The analysis was per protocol.
Measure: Number; unit: participants
Arm/Group | Group A : 40ml Prilocaine 1% | Group B : 30ml Prilocaine 1% | Group C : 20ml Prilocaine 1%
Number analyzed (Participants) | 40 | 40 | 40
participants | 38 | 36 | 32
Statistical Analysis 1: Comparison: Group A : 40ml Prilocaine 1% vs Group B : 30ml Prilocaine 1%; Test type: Superiority or Other; p = 0.675, Fisher Exact
Statistical Analysis 2: Comparison: Group A : 40ml Prilocaine 1% vs Group C : 20ml Prilocaine 1%; Test type: Superiority or Other; p = 0.087, Fisher Exact
Statistical Analysis 3: Comparison: Group B : 30ml Prilocaine 1% vs Group C : 20ml Prilocaine 1%; Test type: Superiority or Other; p = 0.348, Fisher Exact

5. Primary Outcome: Onset Time.
Description: Time from beginning of administration of the local anesthetic until complete sensoric block.
Time Frame: within 60 minutes after administration of the local anesthetic
Population: In some cases the investigators were not able to exactly determine an onset time, so in cases of block failure (supplementation needed) or emergency situations outside this study (onset time not examined). Therefore the number of participants analyzed concerning onset time is lower then the total number of outpatients in each group.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group A : 40ml Prilocaine 1% | Group B : 30ml Prilocaine 1% | Group C : 20ml Prilocaine 1%
Number analyzed (Participants) | 35 | 36 | 36
minutes | 18 (7) | 20 (8) | 26 (10)
Statistical Analysis 1: Comparison: Group A : 40ml Prilocaine 1% vs Group B : 30ml Prilocaine 1%; Test type: Superiority or Other; p = 0.247, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group A : 40ml Prilocaine 1% vs Group C : 20ml Prilocaine 1%; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Group B : 30ml Prilocaine 1% vs Group C : 20ml Prilocaine 1%; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Number of Participants With Subjective Adverse Events as a Measure of Safety and Tolerability.
Description: In groups A, B and C was determined the rate of subjective clinical signs of increased Met-Hb-Levels : headaches or dizziness, when correlated with the peak-Met-Hb-Level.
Time Frame: Outpatients were followed for the duration of hospital stay, an average of six hours.
Measure: Number; unit: participants
Arm/Group | Group A : 40ml Prilocaine 1% | Group B : 30ml Prilocaine 1% | Group C : 20ml Prilocaine 1%
Number analyzed (Participants) | 40 | 40 | 40
participants | 4 | 0 | 0
Statistical Analysis 1: Comparison: Group A : 40ml Prilocaine 1% vs Group B : 30ml Prilocaine 1%; Test type: Superiority or Other; p = 0.116, Fisher Exact
Statistical Analysis 2: Comparison: Group A : 40ml Prilocaine 1% vs Group C : 20ml Prilocaine 1%; Test type: Superiority or Other; p = 0.116, Fisher Exact
Statistical Analysis 3: Comparison: Group B : 30ml Prilocaine 1% vs Group C : 20ml Prilocaine 1%; Test type: Superiority or Other; p = 1, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Group A : 40ml Prilocaine 1% | Group B : 30ml Prilocaine 1% | Group C : 20ml Prilocaine 1%
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 14/40 | 5/40 | 1/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A : 40ml Prilocaine 1% (N=40) | Group B : 30ml Prilocaine 1% (N=40) | Group C : 20ml Prilocaine 1% (N=40)
dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) — Related to regional anesthesia when occuring during the peak of Met-Hb-formation.
headaches (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Related to regional anesthesia when occuring during the peak of Met-Hb-formation.
objective signs of methemoglobinemia (Blood and lymphatic system disorders) | 13 (19) | 5 (5) | 1 (1) — As objective signs of increased concentration of methemoglobin we registrated lip cyanosis and/or drops in oxygen concentration measured with an standard two-wavelength-pulseoximeter.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No